CLINICAL TRIAL: NCT04626180
Title: Effects of Pre-extubation Manual Hyper Inflation in Comparison to Regular Extubation Following Sternotomy.
Brief Title: EFFECT OF PRE EXTUBATION MANUAL HYPERINFLATION TECHNIQUE VS REGULAR EXTUBATION AFTER STERNOTOMY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUI/CTR/2020/7
Record Dates: First submitted 2020-09-18; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-09

CONDITIONS: Sternotomy
Keywords: Sternotomy; Extubation; Manual Hyperinflation
MeSH Terms: interventions — Airway Extubation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular Extubation (Active Comparator)
  Interventions: Procedure: Extubation
- Pre Extubation Manual Hyperinflation (Experimental)
  Interventions: Procedure: Extubation; Procedure: Manual Hyperinflation

INTERVENTIONS:
Procedure: Extubation — Extubation is the removal of an endotracheal tube (ETT), which is the last step in liberating a patient from the mechanical ventilator.
Procedure: Manual Hyperinflation — Providing a larger tidal volume than baseline tidal volume to the patient and using a tidal volume which is 50% greater than that delivered by the ventilator
  Arms: Pre Extubation Manual Hyperinflation

SUMMARY:
Post operative pulmonary complication (PPC) is one of the cause of mortality and morbidity after sternotomy. There is no accessible confirmation which shows the impact of Pre Extubation Manual Hyperinflation method with Regular Extubation procedure. After sternotomy manual hyperinflation technique is not taken during extubation. The objective of the study was to determine the effect of Pre Extubation Manual Hyperinflation technique VS regular Extubation technique on vitals and respiratory parameters in patients after Sternotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 to 60
2. Patient undergone surgery (sternotomy)
3. Elective intubated (ETT orally)
4. Ventilated more than 3 hours -

Exclusion Criteria:

1. Patient with any neurological issue (mentally disturbed) who cannot understand the command
2. Complicated extubation
3. Pulmonary pathology where lung hyperinflation was contra-indicated (e.g. acute respiratory distress syndrome, undrained pneumothorax or exacerbation of chronic obstructive pulmonary disease and acute pulmonary edema.
4. Raised intracranial pressure
5. Redo or reopen. -

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow rate | 1 day
Blood pH | 1 day
Blood pO2 | 1 day
Blood pCO2 | 1 day
Blood pHCO3 | 1 day
Pulse rate | 1 day
Oxygen saturation | 1 day
Forced expiratory volume | 1 day
Forced vital capacity | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria International Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No